CLINICAL TRIAL: NCT06554067
Title: Effects of tDCS and VNS on Postoperative Analgesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Paul Garcia, Associate Professor of Anesthesiology, Division Chief of Neuroanesthesia, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAV2033
Record Dates: First submitted 2024-07-11; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Acute Postoperative Pain
Keywords: Postoperative pain; Chronic Pain; Transcranial direct current stimulation; Vagus nerve stimulation
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This is a parallel-group, double blinded, randomized trial where 200 subjects will be randomized following a 2x2 structure.
Who Masked: Participant, Investigator
Masking Description: Patients will be assigned a Study ID that will determine the assigned procedure. At the study's completion the blind will be broken, and data will be turned over for analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Group +/+ (Experimental): Group +/+ will receive ten minutes of active tDCS followed by ten minutes of active VNS.
  Interventions: Device: Active transcranial direct current stimulation; Device: Active vagus nerve stimulation
- Group +/- (Active Comparator): Group +/- will receive ten minutes of active tDCS followed by ten minutes of sham VNS.
  Interventions: Device: Active transcranial direct current stimulation; Other: Sham vagus nerve stimulation
- Group -/+ (Active Comparator): Group -/+ will receive ten minutes of sham tDCS followed by ten minutes of active VNS.
  Interventions: Device: Active vagus nerve stimulation; Other: Sham transcranial direct current stimulation
- Group -/- (Sham Comparator): Group -/- will receive ten minutes of sham tDCS followed by ten minutes of sham VNS.
  Interventions: Other: Sham transcranial direct current stimulation; Other: Sham vagus nerve stimulation

INTERVENTIONS:
Device: Active transcranial direct current stimulation — Ten minutes of active transcranial direct current stimulation
  Other Names: tDCS
  Arms: Group +/+; Group +/-
Device: Active vagus nerve stimulation — Ten minutes of active vagus nerve stimulation
  Other Names: VNS
  Arms: Group +/+; Group -/+
Other: Sham transcranial direct current stimulation — Ten minutes of sham tDCS
  Arms: Group -/+; Group -/-
Other: Sham vagus nerve stimulation — Ten minutes of sham VNS
  Arms: Group +/-; Group -/-

SUMMARY:
This study seeks to evaluate the efficacy of transcranial direct current stimulation (tDCS) and Afferent Vagus nerve simulation (VNS) in treating acute postoperative pain of patients in the post-anesthesia care unit after general surgery.

Study outcomes will include changes in pain levels and vital signs. For patients who are admitted after surgery, opioid consumption in the 24 hours after surgery and time from surgery to discharge are recorded as secondary outcomes.

Patients will be divided in the following comparison groups:

* Group +/+ will receive ten minutes of active tDCS followed by ten minutes of active VNS.
* Group +/- will receive ten minutes of active tDCS followed by ten minutes of sham VNS.
* Group -/+ will receive ten minutes of sham tDCS followed by ten minutes of active VNS.
* Group -/- will receive ten minutes of sham tDCS followed by ten minutes of sham VNS.

DETAILED DESCRIPTION:
Two nonpharmacologic interventions have shown promise in treatment of chronic pain. Afferent Vagus nerve simulation (VNS) can modulate nociception, even though the exact mechanism is unclear. Clinically, it has found uses in chronic pain as well as early evidence of potential use in postoperative pain. Alternatively, transcranial direct current stimulation (tDCS) is a form of non-invasive and polarity-specific technique of modulating neuronal circuitry using a weak electric current delivered by a battery. tDCS has also been shown to modulate chronic pain and has been shown to produce EEG signatures similar to those seen in states of adequate intraoperative analgesia.

This study seeks to evaluate the efficacy of tDCS and VNS in treating acute postoperative pain of patients in the post-anesthesia care unit after general surgery by randomizing 200 subjects in 4 groups:

* Group +/+ will receive ten minutes of active tDCS followed by ten minutes of active VNS.
* Group +/- will receive ten minutes of active tDCS followed by ten minutes of sham VNS.
* Group -/+ will receive ten minutes of sham tDCS followed by ten minutes of active VNS.
* Group -/- will receive ten minutes of sham tDCS followed by ten minutes of sham VNS.

Patient's vital signs and pain level will be obtained before the procedure and after. Patients that have to stay in hospital will also be evaluated by opioid consumption and time from surgery to discharge.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or above with the capacity to provide informed consent who are undergoing an elective surgery requiring general anesthesia

Exclusion Criteria:

* cardiac bradyarrhythmia: taking beta-blockers;
* patients with metal implants around the chest, neck, or head (e.g. implantable pacemakers and defibrillators, deep brain stimulation devices);
* pregnancy
* history of epilepsy or seizures.
* patients undergoing surgical procedures involving the head, neck or spine, or those requiring the use of cardiopulmonary bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Pain levels using Numerical Rating Scale | Immediately before the intervention and immediately after the intervention.
  Numerical Rating Scale (NRS) from 0-10. 0 being no pain, and 10 being the worse pain patient has experienced.
Pain levels using the Verbal Rating Scale | Immediately before the intervention and immediately after the intervention.
  Verbal Rating Scale (VRS) distinguishing between no pain, mild pain, moderate pain, and severe pain.

SECONDARY OUTCOMES:
Vital Signs: Blood pressure. | Immediately before and immediately after intervention. Then, every 5 minutes until one hour after the intervention.
  Patients at the PACU are under continuous monitoring of vital signs. We will collect the values of the blood pressure in mmHg. A high score (higher than 130/80) will indicate a bad outcome.
Vital Signs: Heart rate | Immediately before and immediately after intervention. Then, every 5 minutes until one hour after the intervention.
  Patients at the PACU are under continuous monitoring of vital signs. We will collect the values of the heart rate before the intervention and after. A result higher than what is physiologic normal (100) will indicate a bad outcome.
Opioid consumption | 24 hours after surgery
  Patients that stay in hospital after surgery will be evaluated for opioid consumption from medical record.
Time from surgery to discharge | From the date of the patient's surgery until the day of the discharge, up to 2 month.
  Investigator will measure how long does the patient stay in the hospital after surgery in number of days.

IPD SHARING:
Plan to Share IPD: No
Data will be shared in aggregate form. There is no plan to share individual participant data (IPD) with researchers not involved with the study design. Several posthoc analyses are being planned for retrospective analysis of the data obtained.